CLINICAL TRIAL: NCT06992752
Title: Investigation of the Properties of Dysfunctional Breathing in Individuals With Thoracic Outlet Syndrome
Brief Title: Dysfunctional Breathing in Individuals With Thoracic Outlet Syndrome
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Melda Saglam, Professor, Hacettepe University
Other Study IDs: SBA-24/775
Record Dates: First submitted 2025-04-29; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Thoracic Outlet Syndrome
Keywords: Thoracic Outlet Syndrome; Dysfunctional Breathing
MeSH Terms: conditions — Thoracic Outlet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thoracic Outlet Syndrome: Thoracic Outlet Syndrome
- Healthy control: Healthy control

SUMMARY:
The aim of this observational study was to learn about the characteristics of dysfunctional breathing in individuals with thoracic outlet syndrome. The main question to be answered is:

Is there a dysfunctional breathing pattern in individuals with Thoracic outlet syndrome? These features will be compared with a healthy control group to evaluate the association of Thoracic outlet syndrome with dysfunctional breathing

ELIGIBILITY:
Inclusion Criteria:

* To agree to participate in the study,
* To have been diagnosed with TOS by a thoracic surgeon,
* To be between 18-65 years old,
* Having pain for more than 6 months

Exclusion Criteria:

* Patients with a history of spinal or thoracic surgery for TOS or any other reason,
* People with traumatic cervical injury,
* Severely obese people (BMI >40 kg/m2),
* People with clinical abnormalities in the thoracic cage or vertebral column,
* Persons with occupational industrial exposures,
* Patients with severe comorbidities (neurological, neuromuscular, -cardiorespiratory, psychiatric and musculoskeletal) diabetes mellitus and/or malignancies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the study, adult patients aged between 18-65 years who were diagnosed with TOS by a thoracic surgeon at the Cardiopulmonary Rehabilitation Unit of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Hacettepe University, and who had pain complaints for more than 6 months without surgery will be evaluated. Control cases planned to be included in the study to compare with the results of the patients will be formed by using the snowball method from the immediate environment.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2025-10-02 (Estimated)

PRIMARY OUTCOMES:
Nijmegen Questionnaire | Day 1
  A cut-off score of ≥20 in Nijmegen will be used to define dysfunctional breathing. The minimum score is 0 and the maximum score is 60 points. Higher scores mean worse outcome.
End tidal CO2 | Day 1
  A standard value of <35 mmHg will be used as the cut-off point for dysfunction
Manual Assessment of Respiratory Motion | 5 minutes
  This technique is used to assess and measure the distribution of respiratory movement between the upper and lower parts of the rib cage and abdomen

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | Day 1
  Forced Vital Capacity (FVC) will be done with a spirometer according to the American Thoracic Society and European Respiratory Society criteria. The total amount of air (L) that can be forced out after taking a deep breath will be recorded. Measures lung capacity.
Forced Expiratory Volume in 1 second (FEV1) | Day 1
  Forced Expiratory Volume in 1 second (FEV1) will be done with a spirometer according to the American Thoracic Society and European Respiratory Society criteria. The amount of air (L) a person can forcefully expel in the first second of a breath will be recorded
FEV1/FVC Ratio | Day 1
  The percentage of the ratio of FEV1 to FVC will be calculated and recorded
Forced Expiratory Flow 25-75% (FEF25-75) | Day 1
  Forced Expiratory Flow 25-75% (FEF25-75%) will be assessed with a spirometer according to American Thoracic Society and European Respiratory Society criteria. The air flow rate (L/s) during the middle part of the exhalation (25%-75%) will be recorded.
Peak Expiratory Flow (PEF) | Day 1
  Peak Expiratory Flow (PEF) will be assessed with a spirometer according to American Thoracic Society and European Respiratory Society criteria. The highest flow rate (L/s) achieved during a forceful exhalation will be recorded.
Breath Holding at Functional Residual Capasity | 5 minutes
  If the duration is less than 25 seconds, it is considered as possible dysfunctional breathing
Breath Holding at Total Lung Capacity | 5 minutes
  If the duration is less than 35 seconds, it is considered as possible dysfunctional breathing
Pain severity | 5 minutes
  Visual analog scale (VAS) will be used in the assessment.Individuals' pain at rest, during activity and at night will be assessed on a scale of 0-10.Minimum score is 0 and maximum score is 10 Higher scores mean a worse outcome.
Pain treshold | 10 minutes
  For the assessment of pain threshold, the minimum pressure value that causes pain or discomfort will be recorded
Pain tolerance | 10 minutes
  the maximum tolerated pressure value will be recorded in the assessment of pain tolerance
Beck Anxiety Scale | 5 minutes
  The scale has 21 questions. The questions will be answered by selecting one of four options: none, mild, moderate and severe. 8-15 points will be categorized as mild anxiety symptoms, 16-25 points as moderate anxiety symptoms, 26 - 63 points as severe anxiety symptoms. the maximum score of the scale is 63
EQ-5D-5L General Quality of Life Scale | 5 minutes
  The scale has two parts. The first section has five sub-scales: movement, self-care, usual activities, pain/discomfort and anxiety/depression. The answers given in each section have 5 options; "no problem", "mild problem", "moderate problem", "severe problem" and "extreme problem". In the second section, individuals give a value between 0 and 100 about their current health status.
Type D Personality Scale | 5 minutes
  It consists of a total of 14 items and two subscales measuring negative affectivity and social inhibition. Each item is scored on a 0-4 scale. The cut-off point of the two subscales is ≥ 10.

CONTACTS AND LOCATIONS:
Overall Officials: Melda Sağlam, Professor, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
for patient data privacy